CLINICAL TRIAL: NCT03483623
Title: NATO Litter: Fluid Immersion System (FIS) Versus Traditional Mattress for Pressure Dispersion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laurie Migliore, Chief, Nursing Research, David Grant U.S. Air Force Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: FDG20160005H
Record Dates: First submitted 2018-03-21; First posted 2018-03-30 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Pressure Distribution; Military Litters; Peak Pressure Index; Total Surface Area; Tissue Perfusion
Keywords: NATO Litter; Dolphin Fluid Immersion System; Raven 90C litter; Transcutaneous oxygenation; WELP mattress

STUDY DESIGN:
Intervention Model Description: This protocol is a Quasi Experimental Cross Factor study. The subject sample is nonrandomized. Subjects will be their own control and have repeated measurements to compare baseline and supine transcutaneous oxygenation levels on four different surface combinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NATO WELP combination (Experimental): Subjects will be their own control and have repeated measurements to compare baseline and supine transcutaneous oxygenation levels and interface pressures on NATO litter and WELP mattress combination
  Interventions: Other: NATO WELP combination
- NATO FIS combination (Experimental): Subjects will be their own control and have repeated measurements to compare baseline and supine transcutaneous oxygenation levels and interface pressures on NATO litter and Fluid Immersion System (FIS) mattress combination
  Interventions: Other: NATO FIS combination
- RAVEN WELP combination (Experimental): Subjects will be their own control and have repeated measurements to compare baseline and supine transcutaneous oxygenation levels and interface pressures on Raven 90C litter and WELP mattress combination
  Interventions: Other: RAVEN WELP combination
- RAVEN FIS combination (Experimental): Subjects will be their own control and have repeated measurements to compare baseline and supine transcutaneous oxygenation levels and interface pressures on Raven 90C litter and Fluid Immersion System (FIS) mattress combination
  Interventions: Other: RAVEN FIS combination

INTERVENTIONS:
Other: NATO WELP combination — Interface pressure will be measured using the XSensor X3 Pressure Mapping System. Transducers will be placed near both scapula. Measures will be obtained in upright (baseline) and supine positions on 4 randomly assigned litter mattress combinations. Constant TCPO2 measures, as well as peak pressures and total body surface area exposed to skin will be measured for the occiput, sacrum, both scapula, buttocks and heel areas. It will take about 20 minutes for each combination. The session is complete after all measures have been obtain for all litter/mattress combinations.
  Arms: NATO WELP combination
Other: NATO FIS combination — Interface pressure will be measured using the XSensor X3 Pressure Mapping System. Transducers will be placed near both scapula. Measures will be obtained in upright (baseline) and supine positions on 4 randomly assigned litter mattress combinations. Constant TCPO2 measures, as well as peak pressures and total body surface area exposed to skin will be measured for the occiput, sacrum, both scapula, buttocks and heel areas. It will take about 20 minutes for each combination. The session is complete after all measures have been obtain for all litter/mattress combinations.
  Arms: NATO FIS combination
Other: RAVEN WELP combination — Interface pressure will be measured using the XSensor X3 Pressure Mapping System. Transducers will be placed near both scapula. Measures will be obtained in upright (baseline) and supine positions on 4 randomly assigned litter mattress combinations. Constant TCPO2 measures, as well as peak pressures and total body surface area exposed to skin will be measured for the occiput, sacrum, both scapula, buttocks and heel areas. It will take about 20 minutes for each combination. The session is complete after all measures have been obtain for all litter/mattress combinations.
  Arms: RAVEN WELP combination
Other: RAVEN FIS combination — Interface pressure will be measured using the XSensor X3 Pressure Mapping System. Transducers will be placed near both scapula. Measures will be obtained in upright (baseline) and supine positions on 4 randomly assigned litter mattress combinations. Constant TCPO2 measures, as well as peak pressures and total body surface area exposed to skin will be measured for the occiput, sacrum, both scapula, buttocks and heel areas. It will take about 20 minutes for each combination. The session is complete after all measures have been obtain for all litter/mattress combinations.
  Arms: RAVEN FIS combination

SUMMARY:
The purpose of this study is to measure peak skin interface pressures and the total area of the body exposed to skin interface pressure above 30 mm Hg at different areas of the body in the supine position on two different support surfaces applied to a standard North Atlantic Treaty Organization (NATO) litter (NSN: 6530-01-380-7309) and a Raven 90C Litter (NSN6530-01-432-5114). The support surfaces are the Warrior Evacuation Litter Pad (WELP) and the Dolphin Fluid Immersion Simulation Stretcher System (FIS). These pressure measurements and transcutaneous oxygenation readings will allow us to determine differences between support surfaces.

DETAILED DESCRIPTION:
The purpose of this study is to measure peak skin interface pressures and the total area of the body exposed to skin interface pressure above 30 mm Hg at different areas of the body in the supine position on two different support surfaces applied to a standard North Atlantic Treaty Organization (NATO) litter (NSN: 6530-01-380-7309) and a Raven 90C Litter (NSN6530-01-432-5114). The Raven 90C is the official litter for the U.S. Navy. It is approved for flight on United States Air Force (USAF) aircraft. It can be easily folded for storage and transport to remote settings. The support surfaces are the Warrior Evacuation Litter Pad (WELP) and the Dolphin Fluid Immersion Simulation Stretcher System (FIS). In theory, mattresses that reduce and/or minimize pressure on the capillary bed's perfusion can help reduce pressure related injury such as pressure or decubitus ulcer development. Skin interface pressure measurements using a pressure mapping system and transcutaneous oxygenation readings will allow us to determine these differences between support surfaces. A better understanding of skin interface pressure associated with the litter support surfaces is vital for military nurses to develop and implement preventative interventions to reduce pressure ulcer development in our patients. In addition, this study will provide information to help determine the usefulness and feasibility of incorporating the fluid immersion system (FIS) as a litter support surface.

This research protocol has one major aim:

To determine the difference in the pressure redistribution qualities between the WELP and the Dolphin FIS

There are also two secondary aims:

1. To determine the difference in the pressure redistribution qualities of the WELP when used as the mattress on the NATO litter and Raven litter.
2. To determine the difference in the pressure redistribution qualities of the Dolphin FIS when used as the mattress on the NATO litter and Raven litter.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years with lawful access to Travis Air Force Base (AFB)

Exclusion Criteria:

* Orthopedic or neurological conditions that prevent a subject from lying flat (supine) without any pillows for head, neck, or lumbar support
* Medical conditions (such as an uncontrollable tremor or twitch) that prevent a subject from staying still for the required periods of time (20 minute increments).
* Pregnancy
* Inability to ambulate unassisted, unstable gate (presenting increased fall risk)
* Extremity prosthetics (hand/arm or foot/leg)
* Height greater than 72 inches (6 feet) - exceeds length of the litter & mattress surfaces
* Body weight greater than 300 lbs
* Subjects who find it difficult, uncomfortable or impossible to remain still for the necessary study time durations (20 minute increments) on the relatively narrow litter surfaces will be removed from the study.
* Subject does not speak or understand the English language

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Migliore, PhD, Principal Investigator — David Grant Medical Center; Antoinette Shinn, PhD, Principal Investigator — 59th Medical Wing
Locations (1):
- David Grant Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bale S, Finlay I, Harding KG. Pressure sore prevention in a hospice. J Wound Care. 1995 Nov;4(10):465-8. doi: 10.12968/jowc.1995.4.10.465. PMID 8548573
- [Background] Bridges EJ, Schmelz JO, Mazer S. Skin interface pressure on the NATO litter. Mil Med. 2003 Apr;168(4):280-6. PMID 12733671
- [Background] Hanson DS, Langemo D, Anderson J, Thompson P, Hunter S. Can pressure mapping prevent ulcers? Nursing. 2009 Jun;39(6):50-1. doi: 10.1097/01.NURSE.0000352337.67771.e0. No abstract available. PMID 19474612
- [Background] International review. Pressure ulcer prevention: pressure, shear, friction and microclimate in context. A consensus document. London: Wounds International, 2010
- [Background] Hatzfeld JJ, Dukes S, Bridges E. Chapter 3 innovations in the en route care of combat casualties. Annu Rev Nurs Res. 2014;32:41-62. doi: 10.1891/0739-6686.32.41. PMID 25222537
- [Background] Harada C, Shigematsu T, Hagisawa S. The effect of 10-degree leg elevation and 30-degree head elevation on body displacement and sacral interface pressures over a 2-hour period. J Wound Ostomy Continence Nurs. 2002 May;29(3):143-8. doi: 10.1067/mjw.2002.123645. PMID 12011906
- [Background] Junkin J, Gray M. Are pressure redistribution surfaces or heel protection devices effective for preventing heel pressure ulcers? J Wound Ostomy Continence Nurs. 2009 Nov-Dec;36(6):602-8. doi: 10.1097/WON.0b013e3181be282f. PMID 19920740
- See also: Strykers' Pioneer (TM) pressure redistributing stretcher surface is the ﬁrst of its kind for emergency departments — http://www.stryker.com/stellent/groups/public/documents/web_assest/006430.pdf
- See also: PeriFlux System 5000 (instrument version 1.70-1.79) Extended User Manual — http://www.perimed-instruments.com
- See also: Pressure effects from a military stretcher. J R Army Med Corps — https://www.ncbi.nlm.nih.gov/pubmed/8277476

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: North Atlantic Treaty Organization (NATO) and Warrior Evacuation Litter Pad (WELP); NATO and Fluid Immersion System (FIS) mattress; Raven 90C litter and WELP; Raven 90C and FIS
Groups:
- NATO WELP/ NATO FIS / RAVEN WELP / RAVEN FIS: Subjects will be their own control and have repeated measurements to compare baseline and supine transcutaneous oxygenation levels, laser Doppler pressure units, and interface pressures on NATO / Raven litters and WELP / FIS mattress combinations
  Interface pressure will be measured using the XSensor X3 Pressure Mapping System. Transducers and probes will be placed near both scapula. Measures will be obtained in upright (baseline) and supine positions on 4 randomly assigned litter mattress combinations. Constant TCPO2 and Doppler measures, as well as peak pressures and total body surface area exposed to skin will be measured for the occiput, sacrum, both scapula, buttocks and heel areas. It will take about 20 minutes for each combination. The session is complete after all measures have been obtain for all litter/mattress combinations.
Period: Overall Study
Arm/Group | NATO WELP/ NATO FIS / RAVEN WELP / RAVEN FIS
Started | 44
Started NATO WELP | 44
Completeded NATO WELP | 43 (1 subject was withdrawn after the target of 43 complete sets was achieved)
Started NATO FIS | 44
Completed NATO FIS | 43 (1 subject was withdrawn after the target of 43 complete sets was achieved)
Started RAVEN WELP | 44
Completed RAVEN WELP | 43 (1 subject was withdrawn after the target of 43 complete sets was achieved)
Started RAVEN FIS | 44
Completed RAVEN FIS | 43 (1 subject was withdrawn after the target of 43 complete sets was achieved)
Completed | 43 (1 subject was withdrawn after the target of 43 complete sets was achieved)
Not Completed | 1
Not completed — 43 complete sets achieved | 1

BASELINE CHARACTERISTICS:
Groups:
- North Atlantic Treaty Organization (NATO) and Warrior Evacuati: Subjects will be their own control and have repeated measurements to compare baseline and supine transcutaneous oxygenation levels, laser Doppler pressure units, and interface pressures on NATO / Raven litters and WELP / FIS mattress combinations. Interface pressure will be measured using the XSensor X3 Pressure Mapping System. Transducers and probes will be placed near both scapula. Measures will be obtained in upright (baseline) and supine positions on 4 randomly assigned litter mattress combinations. Constant TCPO2 and Doppler measures, as well as peak pressures and total body surface area exposed to skin will be measured for the occiput, sacrum, both scapula, buttocks and heel areas. It will take about 20 minutes for each combination. The session is complete after all measures have been obtain for all litter/mattress combinations
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19
  African American | 8
  Hispanic/Latino | 8
  Asian | 3
  Native American/Pacific Islander | 3
  Multiracial/Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43
BMI [Count of Participants; unit: Participants]
  <18.5 | 1
  18.5 - 24.9 | 21
  >25 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pressure Redistribution: Peak Pressure Index
Description: Determine the difference in the pressure redistribution qualities between the WELP and the Dolphin FIS when used as mattress on the NATO litter and Raven litter. Pressure redistribution qualities will be measured in mmHg using XSensor X3 pressure mapping technology. To minimize the risk of a faulty sensor or false reading over one sensor, the average of eight cells around the region will be recorded and referred to as the Peak Pressure Index (PPI). Peak interface pressure is the highest average pressure (mm Hg) measured over vulnerable bony prominences (occiput, sacrum, and bilateral scapula, buttocks, and heels) at 0 minutes. PPI will be measured in mm Hg and the mean will be reported
Time Frame: 0 minutes
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
mm Hg
  NATO WELP | 320.63 (23.46222)
  NATO FIS | 264.8107 (18.91339)
  RAVEN WELP | 328.5933 (22.8568)
  RAVEN FIS | 267.1014 (19.66037)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

2. Primary Outcome: Pressure Redistribution: Peak Pressure Index
Description: Determine the difference in the pressure redistribution qualities between the WELP and the Dolphin FIS when used as mattress on the NATO litter and Raven litter. Pressure redistribution qualities will be measured in mmHg using XSensor X3 pressure mapping technology. To minimize the risk of a faulty sensor or false reading over one sensor, the average of eight cells around the region will be recorded and referred to as the Peak Pressure Index (PPI). Peak interface pressure is the highest average pressure (mm Hg) measured over vulnerable bony prominences (occiput, sacrum, and bilateral scapula, buttocks, and heels) at 5 minutes. PPI will be measured in mm Hg and the mean will be reported
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
mm Hg
  NATO WELP | 312.0279 (23.41317)
  NATO FIS | 255.1633 (17.11509)
  RAVEN WELP | 318.78 (26.95208)
  RAVEN FIS | 257.0823 (18.12933)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

3. Primary Outcome: Pressure Redistribution: Peak Pressure Index
Description: Determine the difference in the pressure redistribution qualities between the WELP and the Dolphin FIS when used as mattress on the NATO litter and Raven litter. Pressure redistribution qualities will be measured in mmHg using XSensor X3 pressure mapping technology. To minimize the risk of a faulty sensor or false reading over one sensor, the average of eight cells around the region will be recorded and referred to as the Peak Pressure Index (PPI). Peak interface pressure is the highest average pressure (mm Hg) measured over vulnerable bony prominences (occiput, sacrum, and bilateral scapula, buttocks, and heels) at 10 minutes. PPI will be measured in mm Hg and the mean will be reported
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
mm Hg
  NATO WELP | 306.5656 (22.72959)
  NATO FIS | 251.1965 (17.01875)
  RAVEN WELP | 312.2267 (25.76947)
  RAVEN FIS | 252.4823 (17.06234)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

4. Primary Outcome: Pressure Redistribution: Peak Pressure Index
Description: Determine the difference in the pressure redistribution qualities between the WELP and the Dolphin FIS when used as mattress on the NATO litter and Raven litter. Pressure redistribution qualities will be measured in mmHg using XSensor X3 pressure mapping technology. To minimize the risk of a faulty sensor or false reading over one sensor, the average of eight cells around the region will be recorded and referred to as the Peak Pressure Index (PPI). Peak interface pressure is the highest average pressure (mm Hg) measured over vulnerable bony prominences (occiput, sacrum, and bilateral scapula, buttocks, and heels) at 15 minutes. PPI will be measured in mm Hg and the mean will be reported
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
mm Hg
  NATO WELP | 304.9372 (23.06759)
  NATO FIS | 247.7028 (15.50624)
  RAVEN WELP | 311.5874 (24.86347)
  RAVEN FIS | 248.243 (15.88815)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

5. Primary Outcome: Pressure Redistribution: Total Surface Area (TSA) > 30 mm Hg
Description: Determine the difference in the pressure redistribution qualities between the WELP when used on the NATO litter and Raven litter. Pressure redistribution will be measured over vulnerable bony prominences as total area of body exposed to skin interface pressures exceeding 30 mm Hg while subjects are in the supine position at 0 minutes. This measure will be expressed as cm2 and the mean will be reported
Time Frame: 0 minutes
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
cm2
  NATO WELP | 778.5449 (198.1991)
  NATO FIS | 610.3898 (218.4296)
  RAVEN WELP | 778.5819 (195.4681)
  RAVEN FIS | 589.0567 (229.7783)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

6. Primary Outcome: Pressure Redistribution: Total Surface Area (TSA) > 30 mm Hg
Description: Determine the difference in the pressure redistribution qualities between the WELP when used on the NATO litter and Raven litter. Pressure redistribution will be measured over vulnerable bony prominences as total area of body exposed to skin interface pressures exceeding 30 mm Hg while subjects are in the supine position at 5 minutes. This measure will be expressed as cm2 and the mean will be reported
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
cm2
  NATO WELP | 693.3249 (180.7349)
  NATO FIS | 501.3781 (198.9074)
  RAVEN WELP | 693.353 (179.1237)
  RAVEN FIS | 488.0037 (205.4465)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

7. Primary Outcome: Pressure Redistribution: Total Surface Area (TSA) > 30 mm Hg
Description: Determine the difference in the pressure redistribution qualities between the WELP when used on the NATO litter and Raven litter. Pressure redistribution will be measured over vulnerable bony prominences as total area of body exposed to skin interface pressures exceeding 30 mm Hg while subjects are in the supine position at 10 minutes. This measure will be expressed as cm2 and the mean will be reported
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
cm2
  NATO WELP | 648.0126 (180.7803)
  NATO FIS | 435.3356 (183.7115)
  RAVEN WELP | 648.0142 (169.5882)
  RAVEN FIS | 432.2805 (192.3748)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

8. Primary Outcome: Pressure Redistribution: Total Surface Area (TSA) > 30 mm Hg
Description: Determine the difference in the pressure redistribution qualities between the WELP when used on the NATO litter and Raven litter. Pressure redistribution will be measured over vulnerable bony prominences as total area of body exposed to skin interface pressures exceeding 30 mm Hg while subjects are in the supine position at 15 minutes. This measure will be expressed as cm2 and the mean will be reported
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
Number analyzed (Participants) | 43
cm2
  NATO WELP | 618.6412 (173.1517)
  NATO FIS | 397.21 (170.7791)
  RAVEN WELP | 619.6928 (171.8377)
  RAVEN FIS | 373.2549 (173.9249)
Statistical Analysis 1: Comparison: North Atlantic Treaty Organization (NATO) and Warrior Evacuati; Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS; Test type: Superiority; p = 0.0001, ANOVA — Statistical analysis applies to all combinations-NATO WELP, NATO FIS, RAVEN WELP, RAVEN FIS

ADVERSE EVENTS:
Time Frame: through study completion, up to 2 hours
Arm/Group | North Atlantic Treaty Organization (NATO) and Warrior Evacuati
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03483623/Prot_SAP_000.pdf